CLINICAL TRIAL: NCT02603575
Title: Effects and Safety of Caspofungin and Corticosteroids in Pneumocystis Pneumonia in Non-HIV Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Hangyong He, Doctor, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BeijingCYHRICU01
Record Dates: First submitted 2015-11-08; First posted 2015-11-13 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-01

CONDITIONS: Pneumocystis Pneumonia
Keywords: Caspofungin; corticosteroids; Pneumocystis Pneumonia; Immunocompromised; Non-HIV; respiratory failure
MeSH Terms: conditions — Pneumonia, Pneumocystis; Respiratory Insufficiency | interventions — Caspofungin; Adrenal Cortex Hormones; Methylprednisolone; Sulfanilamides

ARMS (4):
- Caspofungin and corticosteroids (Experimental): patients treat with caspofungin and corticosteroids on the base of sulfanilamide
  Interventions: Drug: caspofungin; Drug: corticosteroids; Drug: Sulfanilamides
- Caspofungin and no corticosteroids (Active Comparator): patients treat with caspofungin on the base of sulfanilamide
  Interventions: Drug: caspofungin; Drug: Sulfanilamides
- corticosteroids and no caspofungin (Active Comparator): patients treat with corticosteroids on the base of sulfanilamide
  Interventions: Drug: corticosteroids; Drug: Sulfanilamides
- no corticosteroids and no caspofungin (Active Comparator): patients treat with sulfanilamide only
  Interventions: Drug: Sulfanilamides

INTERVENTIONS:
Drug: caspofungin — 70mg ivdrip the first day, then 50mg ivdrip qd
  Arms: Caspofungin and corticosteroids; Caspofungin and no corticosteroids
Drug: corticosteroids — 40mg ivdrip q12h for 5 days 40mg ivdrip qd for 5 days 20mg po for 11 days
  Other Names: methylprednisolone
  Arms: Caspofungin and corticosteroids; corticosteroids and no caspofungin
Drug: Sulfanilamides — 1.92g q8h

SUMMARY:
Pneumocystis Pneumonia is increasing in Immunocompromised Non-HIV Infected Patients. The effects and safety of caspofungin and corticosteroids is not certain in this population. All Immunocompromised Non-HIV patients with respiratory failure were randomized into caspofungin and non-caspofungin group and corticosteroids and non-steroids group. The major outcome is 28 day mortality, the second outcome are time of respiratory rate decreases to less than 25 breath per minute, body temperature lower than 37.3℃.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised Non-HIV Infected Patients
* Partial arterial O2 pressure(PaO2)/FiO2≤300mmHg
* Diagnosed as Pneumocystis Pneumonia

Exclusion Criteria:

* younger than 16 years old
* severe organ failure
* allergic to sulfanilamide, caspofungin or corticosteroid

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 days

SECONDARY OUTCOMES:
Time for release of fever | 2 days
  Time for body temperature less than 37.3℃ for 48 hours
Time for release of respiratory distress | 2 days
  Time for respiratory rate <25 breathes per minute for 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao Yang Hospital, Beijing, China